CLINICAL TRIAL: NCT00693069
Title: Effect of Different Dosing Regimens of Clopidogrel Given Before Elective Percutaneous Coronary Intervention on Platelet Function
Brief Title: Effect of Different Dosing Regimens of Clopidogrel Before Elective Percutaneous Coronary Intervention (PCI) on Platelet Function
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Responsible Party: Jean G Diodati, MD, Hopital du Sacre-Coeur de Montreal
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C.E.2004-06-24A
Record Dates: First submitted 2008-06-03; First posted 2008-06-06 (Estimated); Last update posted 2012-08-21 (Estimated); Status verified 2008-06

CONDITIONS: Coronary Artery Disease
Keywords: angioplasty; clopidogrel; coronary artery disease; platelets; Percutaneous coronary intervention
MeSH Terms: conditions — Coronary Artery Disease | interventions — Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): Clopidogrel 300 mg the day before PCI
  Interventions: Drug: Clopidogrel
- 2 (Experimental): Clopidogrel 600 mg the day before PCI
  Interventions: Drug: Clopidogrel
- 3 (Experimental): 300 mg followed by 75 mg daily started one week prior to angiography
  Interventions: Drug: Clopidogrel
- 4 (Experimental): 300 mg followed by 150 mg daily started one week prior to angiography
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — clopidogrel 300 mg on the day prior to angiography
  Arms: 1
Drug: Clopidogrel — clopidogrel 600 mg on the day prior to angiography
  Arms: 2
Drug: Clopidogrel — clopidogrel 300 mg followed by 75 mg daily started one week prior to angiography
  Arms: 3
Drug: Clopidogrel — clopidogrel 300 mg followed by 150 mg daily started one week prior to angiography
  Arms: 4

SUMMARY:
Adequate platelet inhibition before percutaneous coronary intervention (PCI) reduces peri-procedural and long-term ischemic complications. Documented reduced response to clopidogrel has been associated with subsequent major adverse cardiovascular events. Strategies to optimize platelet inhibition pre-PCI are under investigation.

This study sought to evaluate the effect on platelet aggregation of four different dosing regimens of clopidogrel given before elective PCI.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient with an indication for elective coronary angiography with or without PCI

Exclusion Criteria:

* major hemorrhagic diathesis or active bleeding
* acute myocardial infarction (MI) within 14 days of enrolment
* unstable angina with ST-segment changes >1 mm in at least two contiguous electrocardiographic leads at rest or a troponin I level >0.06 microg/L within 14 days of enrolment
* stroke within the past 3 months
* platelet count <100 x 10 9/L
* prothrombin time > 1.5 times control
* hematocrit <25% or hemoglobin level <100 g/L
* alcohol or drug abuse
* enrolment in other investigational drug trials within the previous month
* use of thienopyridines, glycoprotein (GP) IIb/IIIa inhibitors, warfarin or acenocoumarol within the previous week
* allergic reaction or any contraindication to clopidogrel or aspirin administration

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2004-09; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study was to evaluate the effect of four different dosing regimens of clopidogrel on platelet aggregation at the time of diagnostic coronary angiography, and 2 hours after stenting. | 7 days

SECONDARY OUTCOMES:
A secondary objective in patients stented was the 30-day incidence of the composite of death, myocardial infarction (MI) or urgent target vessel revascularization. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Jean G Diodati, MD, Principal Investigator — Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Locations (1):
- Hopital du Sacre-Coeur de Montreal, Montreal, Quebec, Canada